CLINICAL TRIAL: NCT06821711
Title: Targeting LDL-C to Less Than 0.8 mmol/L in Patients After PCI With High Risk of Cardiovascular Disease: an Open-label, Assessor-blinded, Randomized Trial (REC-SAFETARGET Trial)
Brief Title: Optimal LDL-C Target in High-risk Patients After PCI
Acronym: REC-SAFETARGET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor in Cardiology, Director of the Department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20242295-F-1
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Coronary Syndrome; Acute Coronary Syndromes; Percutaneous Coronary Intervention; High Risk Patient
Keywords: Acute coronary syndrome; Chronic coronary syndrome; Percutaneous coronary intervention; LDL-C; lipid
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDL-C target < 0.8 mmol/L (Experimental): After randomization, investigators will optimize the intensive lipid-lowering regimen based on the patient's prior medication history, baseline LDL-C level, and target LDL-C level, adjusting and titrating LDL-C levels to achieve the target range.
  Interventions: Other: Intensive LDL-C control
- LDL-C target of 0.8 to 1.4 mmol/L (Active Comparator): After randomization, investigators will optimize the intensive lipid-lowering regimen based on the patient's prior medication history, baseline LDL-C level, and target LDL-C level, adjusting and titrating LDL-C levels to achieve the target range.
  Interventions: Other: Conventional LDL-C control

INTERVENTIONS:
Other: Intensive LDL-C control — By Statin, Ezetimibe, or PCSK9i, prescribed according to LDL-C level at baseline and follow-up;
  For patients with baseline LDL-C level < 3.0 mmol/L, it is recommended to start lipid control by statin + PCSK9i; for LDL-C level ≥ 3.0 mmol/L, statin + ezetimibe + PCSK9i
  Arms: LDL-C target < 0.8 mmol/L
Other: Conventional LDL-C control — By Statin, Ezetimibe, or PCSK9i, prescribed according to LDL-C level at baseline and follow-up;
  For patients with baseline LDL-C level < 3.0 mmol/L, it is recommended to start lipid control by statin alone or statin + ezetimibe; for LDL-C level ≥ 3.0 mmol/L, statin + PCSK9i
  Arms: LDL-C target of 0.8 to 1.4 mmol/L

SUMMARY:
Extensive evidence from epidemiological, genetic, and randomized controlled trials (RCTs) of lipid-lowering therapies has firmly established a causal relationship between low-density lipoprotein cholesterol (LDL-C) and atherosclerotic cardiovascular disease (ASCVD), establishing LDL-C as both a pathogenic risk factor and a critical therapeutic target.

Lipid-lowering therapies targeting LDL-C have significantly decreased the overall risk in ASCVD patients. Consequently, current guidelines recommend, based on risk stratification, lowering LDL-C levels in high-risk ASCVD patients to <1.4 mmol/L with a ≥50% reduction from baseline. Findings from PROVE IT-TIMI 22, IMPROVE-IT, ODYSSEY OUTCOMES, and FOURIER-OLE trials suggest that achieving extremely low LDL-C levels may further reduce the risk of cardiovascular events in ASCVD patients without substantially increasing clinically relevant adverse events; however, randomized data was still scarce in supporting this notion.

Against these backgrounds, we have designed this trial to investigate whether targeting LDL-C levels <0.8 mmol/L in high-risk ASCVD patients results in a significant reduction in adverse events compared to targeting LDL-C levels of 0.8-1.4 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent percutaneous coronary intervention due to acute or chronic coronary syndrome
2. Patients with ASCVD at extremely high risk
3. Patients who are able to complete the follow-up and compliant with the allocated treatment

   * ASCVD at extremely high risk is defined as fulfilling at least TWO of the following criteria:

     1. PCI for acute myocardial infarction (AMI, including STEMI or NSTEMI)
     2. Previous AMI, previous stroke, or previous intervention or surgery for peripheral vascular disease
     3. Experienced cardiovascular event(s) with LDL-C≤1.8mmol/L
     4. LDL-C≥4.9mmol/L
     5. Diabetes
     6. CKD (eGFR < 60 ml/min/1.73m2)
     7. Current smoking
     8. Recurrent cardio/cerebrovascular events
     9. History of premature ASCVD (< 55 male, < 65 female)
     10. Complex PCI (fulfilling at least one of the following criteria: multivessel disease; in-stent restenosis; ≥ 3 stents implanted; total stent length ≥ 60 mm; bifurcation; left main disease; target lesions allocated in bypass graft; chronic total occlusion (≥ 3 months of occlusion))

Exclusion Criteria:

1. Age less than 18 years;
2. Unable to give informed consent or currently participating in other trials;
3. Patient who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to randomization in women of child-bearing potential according to local practice), or plans to become pregnant during treatment;
4. Concurrent medical condition with a life expectancy of less than 3 years;
5. Hemodynamic unstable;
6. Active liver disease or hepatic dysfunction (persistent unexplained ALT/AST elevations (≥ 3 × ULN)), patients with a transient increase ALT/AST due to the acute MI may be enrolled;
7. Unable to reach the LDL-C target by known intolerance or contradiction of lipid control medications;
8. LDL-C ≤ 1.4 mmol/L at baseline without any lipid control medication lowering LDL-C;
9. Known active infection or critical hematologic/endocrine dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2029-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events | 24 months
  MACCE, a composite of cardiovascular death, stroke, myocardial infarction, and any revascularization.

SECONDARY OUTCOMES:
Patient-oriented composite endpoint | 24 months
  PoCE, a composite of all-cause death, stroke, myocardial infarction, revascularization, is the first major secondary outcome.
Device-oriented Composite Endpoint | 24 months
  DoCE, a composite of cardiovascular death, target vessel myocardial infarction, clinically and physiologically-indicated target lesion revascularization, is the second major secondary outcome.
Composite of all-cause death, stroke, and myocardial infarction | 24 months
  The composite of all-cause death, stroke, and myocardial infarction is the third major secondary outcome.
All-cause death | 24 months
  All-cause death is considered as other secondary endpoint
Cardiovascular death | 24 months
  Cardiovascular death is considered as other secondary endpoint
Myocardial infarction | 24 months
  Myocardial infarction is considered as other secondary endpoint
Stroke | 24 months
  Stroke is considered as other secondary endpoint
Ischemic stroke | 24 months
  Ischemic stroke is considered as other secondary endpoint
Hemorrhagic stroke | 24 months
  Hemorrhagic stroke is considered as other secondary endpoint
Revascularization | 24 months
  Revascularization is considered as other secondary endpoint
Target lesion revascularization | 24 months
  Target lesion revascularization is considered as other secondary endpoint
Clinically and physiologically-indicated target lesion revascularization | 24 months
  Clinically and physiologically-indicated target lesion revascularization is considered as other secondary endpoint
Cardiovascular hospitalization | 24 months
  Cardiovascular hospitalization is considered as other secondary endpoint

OTHER OUTCOMES:
EuroQol-5D-5L | 24 months
  EuroQol-5D-5L is considered as exploratory endpoint
Everyday Cognition Questionnaire | 24 months
  Everyday Cognition Questionnaire is considered as exploratory endpoint
Pharmacological costs | 24 months
  Pharmacological costs is considered as exploratory endpoint
All adverse events | 24 months
  All adverse events is defined by CTCAE V5.0, considered as safety endpoint
All serious adverse events | 24 months
  All serious adverse events is defined by CTCAE V5.0, considered as safety endpoint
Adverse events of interest | 24 months
  Adverse events of interest, including minor bleeding, major bleeding, injection site reactions, allergic reactions, muscle-related adverse events, rhabdomyolysis, cataracts, adjudicated case of new-onset diabetes, neurocognitive disorders, AST/ALT elevation >3 times the upper limit of normal, creatine kinase elevation >5 times the upper limit of normal, which is considered as safety endpoint
  Adverse events of interest is the safety endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, Ph.D., M.D., Study Chair — Department of Cardiology, Xijing Hospital; Chao Gao, Ph.D., M.D., Study Chair — Department of Cardiology, Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No